CLINICAL TRIAL: NCT03738696
Title: Efficacy of Liposomal Bupivacaine in Arthroscopic Rotator Cuff Repair
Brief Title: Liposomal Bupivacaine in Rotator Cuff Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Amit Momaya, Associate Professor, Orthopaedic Surgery, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002544
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Rotator Cuff Injury
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal bupivacaine Interscalene Block (Experimental): Interscalene block:
  * 10cc (133mg) liposomal bupivacaine;PLUS
  * 10cc 0.25% bupivacaine
  Interventions: Drug: Exparel
- Ropivacaine Interscalene Catheter (Active Comparator): * 20cc 0.25% bupivacaine interscalene block; PLUS
  * Ropivacaine 0.25% interscalene catheter (6ml/hr for 48hrs)
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Exparel — A long-acting injectable sodium channel blocker bound to lipid that is indicated in controlling postoperative pain
  Other Names: liposomal bupivacaine
  Arms: Liposomal bupivacaine Interscalene Block
Drug: Ropivacaine — A short-acting injectable sodium channel blocker bound to lipid that is indicated in controlling postoperative pain
  Arms: Ropivacaine Interscalene Catheter

SUMMARY:
To assess the efficacy of interscalene liposomal bupivacaine in controlling postoperative pain scores, oral morphine equivalents and sleep quality after arthroscopic rotator cuff repair surgery as compared to interscalene catheter.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing outpatient arthroscopic rotator cuff repair
* Greater than or equal to 19 years of age at the time of surgery

Exclusion Criteria:

* Planned operative fixation of the biceps tendon or acromioclavicular joint
* Opioid use 6 weeks before surgery
* Gabapentin use 6 weeks before surgery
* History of prior shoulder surgery on the operative limb
* Severe pulmonary dysfunction
* Diagnosis of chronic pain, fibromyalgia or other somatosensory disorder(s)
* History of radicular pain or neuropathy in the operative limb
* Patients who are currently incapacitated for medical decision making

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UAB Hospital-Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine Block: 10 mL (133 mg) of liposomal bupivacaine mixed with 7 mL (35 mg) bolus of 0.5% bupivacaine
  Exparel: A long-acting injectable sodium channel blocker bound to lipid that is indicated in controlling postoperative pain
- Ropivacaine Interscalene Catheter: * bolus of 15-20 mL of 0.5% ropivacaine given through the needle prior to threading the catheter
  * 0.2% ropivacaine started in the post-anesthesia care unit at 8 mL/hour for 48 hours
  Ropivacaine: A short-acting injectable sodium channel blocker bound to lipid that is indicated in controlling postoperative pain
Period: Overall Study
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Started | 28 | 36 (On the morning of surgery, one patient who was randomized to the ISC arm withdrew from the study without undergoing intervention)
Completed | 20 | 21
Not Completed | 8 | 15
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 8 | 14

BASELINE CHARACTERISTICS:
Population: One patient that was randomized to ropivacaine interscalene catheter arm withdrew from the study prior to intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter | Total
Number analyzed (Participants) | 28 | 35 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.9) | 54.2 (13.0) | 55.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 17 | 21 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 35 | 63
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 31.8 (6.8) | 33.0 (5.8) | 32.5 (6.2)
Tobacco Use [Number; unit: participants] | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Average Postoperative Pain Scores Over a 96 Hour Timeframe
Description: Visual analog pain scores after operation [0-10, with 10 being the worst pain]
Time Frame: Up to 96 hrs postoperative
Population: In the 96 hour timeframe, only 33 of the 35 patients in the Ropivacaine Interscalene Catheter group filled out their surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Number analyzed (Participants) | 28 | 33
score on a scale | 3.0 (2.7) | 3.5 (3.0)

2. Secondary Outcome: Average Postoperative Oral Morphine Equivalents Over a 96 Hour Timeframe
Description: oral morphine equivalents of all opioid-containing medications received
Time Frame: Up to 96 hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Number analyzed (Participants) | 28 | 33
morphine milligram equivalents | 56.4 (42.9) | 58.5 (40.8)

3. Secondary Outcome: Average Analgesia Satisfaction Over a 96 Hour Timeframe
Description: Likert scale of analgesia satisfaction [0-5, with 5 being the most satisfied]
Time Frame: Up to 96 hrs
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Number analyzed (Participants) | 28 | 33
score on a scale | 4.4 (0.9) | 4.4 (0.8)

4. Secondary Outcome: Percentage of Participants With Analgesia Complications
Description: Complications resulting from the method of analgesia utilized
Time Frame: Up to 96 hrs
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Number analyzed (Participants) | 28 | 33
percentage of participants | 13.1 | 29.8

5. Secondary Outcome: Average Sleep Quality Over a 96 Hour Timeframe
Description: Scale of sleep quality [0-10, with 10 being the most satisfied]
Time Frame: Up to 96 hrs postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Number analyzed (Participants) | 28 | 33
score on a scale | 5.7 (2.5) | 5.2 (2.6)

6. Secondary Outcome: Average Hours of Painless Sleep
Description: Hours of sleep uninterrupted by pain [numerical, hours]
Time Frame: Up to 96 hrs postoperative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours of uninterrupted sleep (longest)
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
Number analyzed (Participants) | 28 | 33
hours of uninterrupted sleep (longest) | 4.9 (2.5) | 4.4 (2.4)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Liposomal Bupivacaine Block | Ropivacaine Interscalene Catheter
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/33
Other Adverse Events (participants affected / at risk) | 8/28 | 12/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine Block (N=28) | Ropivacaine Interscalene Catheter (N=33)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT03738696/Prot_SAP_001.pdf